CLINICAL TRIAL: NCT02680951
Title: Dasatinib in Combination With Chemotherapy for Relapsed or Refractory Core Binding Factor Acute Myeloid Leukemia: A Phase I Study (AflacLL1401)
Brief Title: Dasatinib in Combination With Chemotherapy for Relapsed or Refractory Core Binding Factor Acute Myeloid Leukemia
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: Withdrawn due to lack of participants.
Sponsor: Emory University (Other)
Responsible Party: Principal Investigator, Melinda Pauly, MD, Emory University
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB00078620
Record Dates: First submitted 2016-02-09; First posted 2016-02-12 (Estimated); Last update posted 2018-04-19 (Actual); Status verified 2018-04

CONDITIONS: Acute Myeloid Leukemia
Keywords: Pediatric; Adolescent
MeSH Terms: conditions — Leukemia, Myeloid, Acute | interventions — Dasatinib; fludarabine; fludarabine phosphate; Cytarabine; Idarubicin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Dose Level 1 (Experimental): Study participants #1 - #6 receive dose level 1 of dasatinib (60/mg/m2/day) in addition to the standard treatment, for up to 2 courses. Each treatment course is 29 days.
  Treatment course 1 consists of:
  * Fludarabine at a dose of 30mg/m2, intravenously once daily on days 1-5
  * Cytarabine at a dose of 2000mg/m2, intravenously once daily on days 1-5
  * Idarubicin at a dose of 8mg/m2, intravenously once daily on days 3-5
  * Intrathecal cytarabine on day 1 according to standard age specific dosing guidelines
  * Dasatinib orally, once daily on days 6-29
  Participants achieving a response of standard disease or better are eligible for course 2 consisting of dasatinib with fludarabine and cytarabine alone.
  Interventions: Drug: Dasatinib; Drug: Fludarabine; Drug: Cytarabine; Drug: Idarubicin; Drug: Intrathecal (IT) cytarabine
- Dose Level 2 (Experimental): Study participants # 7 - # 12 receive dose level 2 of dasatinib (80/mg/m2/day) in addition to the standard treatment (up to 2 courses), if the participants receiving Dose Level 1 did not experience intolerable side effects. Each treatment course is 29 days.
  Treatment course 1 consists of:
  * Fludarabine at a dose of 30mg/m2, intravenously once daily on days 1-5
  * Cytarabine at a dose of 2000mg/m2, intravenously once daily on days 1-5
  * Idarubicin at a dose of 8mg/m2, intravenously once daily on days 3-5
  * Intrathecal cytarabine on day 1 according to standard age specific dosing guidelines
  * Dasatinib orally, once daily on days 6-29
  Participants achieving a response of standard disease or better are eligible for course 2 consisting of dasatinib with fludarabine and cytarabine alone.
  Interventions: Drug: Dasatinib; Drug: Fludarabine; Drug: Cytarabine; Drug: Idarubicin; Drug: Intrathecal (IT) cytarabine
- Dose Level 3 (Experimental): Study participants # 13 - # 18 receive dose level 3 of dasatinib (100/mg/m2/day) in addition to the standard treatment (up to 2 courses), if the participants receiving Dose Level 2 did not experience intolerable side effects. Each treatment course is 29 days.
  Treatment course 1 consists of:
  * Fludarabine at a dose of 30mg/m2, intravenously once daily on days 1-5
  * Cytarabine at a dose of 2000mg/m2, intravenously once daily on days 1-5
  * Idarubicin at a dose of 8mg/m2, intravenously once daily on days 3-5
  * Intrathecal cytarabine on day 1 according to standard age specific dosing guidelines
  * Dasatinib orally, once daily on days 6-29
  Participants achieving a response of standard disease or better are eligible for course 2 consisting of dasatinib with fludarabine and cytarabine alone.
  Interventions: Drug: Dasatinib; Drug: Fludarabine; Drug: Cytarabine; Drug: Idarubicin; Drug: Intrathecal (IT) cytarabine

INTERVENTIONS:
Drug: Dasatinib — Administered orally on a once daily schedule based on the dose level assigned to the patient at enrollment (60, 80, or 100mg/m2/day). Patients may adjust the time they take dasatinib as long as they take the drug approximately every 24 hours
  Other Names: Sprycel; BMS-354825
Drug: Fludarabine — 30 mg/m2/dose, intravenous infusion over 30 minutes, once daily, on days 1 to 5, total 5 doses
  Participants with body weight less than 12Kg, the fludarabine dose will be corrected as follows: [weight (Kg) x dose (per m2)] divided by 30
  Other Names: Fludara
Drug: Cytarabine — 2000 mg/m2/dose intravenous infusion over 1 to 3 hours, starting 4 hours after the beginning of fludarabine, once daily, on days 1 to 5, total 5 doses
  Participants with body weight less than 12Kg, the cytarabine dose will be corrected as follows: [weight (Kg) x dose (per m2)] divided by 30
  Other Names: Depocyt; Cytosar-U
Drug: Idarubicin — 8mg/m2/dose intravenous infusion over 15 minutes, once daily, on days 3 to 5, total 3 doses
  Participants with body weight less than 12Kg, the idarubicin dose will be corrected as follows: [weight (Kg) x dose (per m2)] divided by 30
  Other Names: Idamycin
Drug: Intrathecal (IT) cytarabine — Given intrathecally to all participants on day 1 of course 1 and 2. Omit on day 1 of course 1 if participant received IT therapy within 7 days prior to study enrollment. Intrathecal chemotherapy may be given during the end of course 1 disease evaluation (spinal fluid and bone marrow aspiration) and may be repeated every 7 days with bone marrow evaluations per institutional preference.
  Cytarabine dose defined by age:
  * 30 mg for patients age 1 - 1.99
  * 50 mg for patients age 2 - 2.99
  * 70 mg for patients ≥3 years of age
  The participant may receive intrathecal triple therapy (ITT) if persistent blasts are present in the cerebral spinal fluid (CSF) based on the treating physician's clinical judgment.
  Other Names: Depocyt; Cytosar-U

SUMMARY:
This study will examine the appropriate dose and side effects of dasatinib, when it is given with the standard of care chemotherapy for children and adolescents with Acute Myeloid Leukemia (AML).

DETAILED DESCRIPTION:
This Phase I study is for children and adolescents who have acute myelogenous leukemia (AML) that has come back (relapsed) or has become resistant (refractory) to standard therapies. Researchers want to know if a drug called dasatinib is safe when used together with standard chemotherapy in treating patients who have relapsed or have resistant AML. Their leukemia has a particular genetic mutation, called core-binding factor.

This type of leukemia has an increase of a cancer promoting protein called c-KIT. Dasatinib can target this protein in laboratory experiments. Laboratory and other studies suggest that dasatinib may prevent acute myeloid leukemia cells from growing and may lead to the destruction of leukemia cells.

The main goal of this study is to find a safe dose of dasatinib and to find out the side effects of dasatinib when it is given in combination with standard chemotherapy to children and adolescents. Similar studies are currently being done in adult patients. Dasatinib has been proven safe and effective in the treatment of other types of leukemia, both by itself and in combination with standard chemotherapy. It is not, however, FDA-approved for use in children.

Three to six participants will receive the starting dose of the drug. If the side effects are not too severe, the next group of participants will take the study drug at a higher dose level. Up to two dose levels of the study drug will be tested. Dasatinib is given by mouth once daily on days 6 to 29 of each 42-day cycle. Participants may receive two cycles in this study.

In addition to dasatinib, participants receive chemotherapy intravenously (IV) with fludarabine, cytarabine, idarubicin, as well as in the spinal fluid (intrathecal or IT chemotherapy). Intrathecal chemotherapy includes cytarabine at the start of each cycle. These drugs are part of standard AML treatment. If at the time of study entry a subject has leukemia cells in their spinal fluid (CNS leukemia), they may receive additional intrathecal chemotherapy with cytarabine, methotrexate, and hydrocortisone (IT triples) during each cycle.

Required research tests include pharmacokinetic (PK) and pharmacodynamics (PD) blood draws (about 1 teaspoon each time) during cycle 1. Optional research tests include extra marrow (about 1 teaspoon each time) for genetic testing and banking of marrow (1 teaspoon) for future studies about cancer.

Primary Objectives of this study are:

* To evaluate the safety of combining dasatinib with reinduction chemotherapy comprised of idarubicin, fludarabine and cytarabine (Ida - FLU/Ara) in children with relapsed or refractory core binding factor acute myeloid leukemia (CBF AML)
* To characterize the toxicity profile of this combination in pediatric patients with relapsed or refractory CBF AML

Secondary Objectives of this study are:

* To estimate the response rates to the combination chemotherapy in the context of a Phase I study, in children with AML in first or greater relapse or refractory to induction chemotherapy
* To determine the genotype of c-KIT exons 8 and 17 and correlate with response rate
* To characterize c-KIT expression of bone marrow blasts at study entry and at the end of course 1 of therapy and describe any correlation with response to therapy

Exploratory Objectives are:

* To investigate descriptively the pharmacodynamic modulation of c-KIT target, Stat3, in a cell line by patient-derived plasma
* To perform RNA sequencing on bone marrow samples at study entry in order to describe the prevalence of mutations in AML associated genes, including c-KIT, and correlate descriptively with progression free survival
* To collect biology specimens at study entry and completion of therapy for future biology studies

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed relapsed or refractory Acute Myeloid Leukemia (AML) and meet the following criteria: Relapsed disease is defined as AML in 1st or greater marrow relapse; Refractory disease is defined as AML which failed to go into remission after 1st or greater relapse, OR AML which failed to go into remission after two or more induction attempts from original diagnosis
* ≥ 5% blasts by morphology in the bone marrow or molecular evidence of at least 0.1% leukemic blasts in the bone marrow
* Definitive evidence of t(8;21) or inv(16) by a CLIA approved cytogenetics laboratory from initial diagnosis
* CNS or other sites of extramedullary disease. No cranial irradiation is allowed during the protocol therapy
* Lansky ≥ 50 for patients ≤ 16 years old; Karnofsky ≥ 50 for patients > 16 years old
* Have fully recovered from the acute toxic effects of all prior chemotherapy, immunotherapy, or radiation therapy prior to entering this study
* Have adequate renal and hepatic functions
* A shortening fraction greater than or equal to 27% by echocardiogram, OR ejection fraction greater than or equal to 50% by radionuclide angiogram (MUGA)
* Must not have any evidence of dyspnea at rest, exercise intolerance, and must have a pulse oximetry > 94% at sea level
* Patients with a seizure disorder may be enrolled if well controlled on anticonvulsants at a dose that has been stable for at least 14 days
* Female participants of childbearing potential must have a negative urine or serum pregnancy test confirmed within 24 hours prior to enrollment
* Female participants with infants must agree not to breastfeed their infants while on this study
* Male and female participants of child-bearing potential must agree to use an effective method of contraception approved by the investigator during the study and for a minimum of 6 months after study treatment

Exclusion Criteria:

* Known allergy to any of the drugs used in the study
* Systemic fungal, bacterial, viral or other infection of which they exhibit ongoing signs/symptoms related to the infection without improvement despite appropriate antibiotics or other treatment
* Any clinically significant cardiovascular disease including: myocardial infarction or ventricular tachyarrhythmia within 6 months, prolonged QTc > 480 msec by the Fridericia correction, major conduction abnormality, such as 2nd or 3rd degree heart block or symptomatic bundle branch block, unless a cardiac pacemaker is present
* Plans to administer non-protocol chemotherapy, radiation therapy, or immunotherapy during the study period
* Refractory to red blood cell or platelet transfusions
* Receiving anti-coagulation therapy
* A need to administer drugs that inhibit platelet function, such as aspirin or clopidogrel
* Receiving any of the following potent CYP3A4 inducers or inhibitors: erythromycin, clarithromycin, ketoconazole, azithromycin, itraconazole, grapefruit juice or St. John's Wort
* Significant concurrent disease, illness, psychiatric disorder or social issue that would compromise patient safety or compliance with the protocol treatment or procedures, interfere with consent, study participation, follow up, or interpretation of study results
* Individuals with Down syndrome and DNA fragility syndromes (such as Fanconi anemia, Bloom syndrome)

Ages: 1 Year to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 0 (Actual)
Dates: Start 2015-12 (Actual); Primary Completion 2017-12-15 (Actual); Study Completion 2017-12-15 (Actual)

PRIMARY OUTCOMES:
Safety of Dasatinib assessed by the Number of Adverse Events | Duration of Study (Up to 161 Days)
  The number of adverse events throughout the duration of the study will be collected to assess the safety of dasatinib.
Number of Dose-Limiting Toxicities (DLT) | Duration of Course 1 (Up to 42 Days)
  The number of dose limiting toxicities (DLT) as defined by grade 3 or higher non-hematologic adverse events persisting for great than 48 hours without resolution to a grade 2 or less, grade 2 pleural effusion that persists longer than 1 week, failure to recover an absolute neutrophil count (ANC) of greater than 500/µL, and platelet count of greater than 50,000/µL. Dose level toxicities will be assessed in the first course only.
Maximum Tolerated Dose (MTD) | Duration of Study (Up to 161 Days)
  The MTD will be the highest dose at which 1 or fewer of six patients experience dose-limiting toxicities (DLT).

SECONDARY OUTCOMES:
Remission Status assessed by Bone Marrow Aspiration/Biopsy | Between Day 29 and Day 43
  A single bone marrow aspiration/biopsy will be performed to assess remission status between day 29 and 43. The exact time point of the bone marrow aspiration/biopsy is dependent on blood count recovery (absolute neutrophil count of greater than 500). Day 43 is the last day remission status must be assessed.
Effect of Dasatinib on c-KIT Expression assessed by Phosphorylation of Stat3 | Baseline, End of course 1 (Up to 49 days)
  The effect of dasatinib on c-KIT expression will be measured by phosphorylation of Stat3 in a core binding factor acute myeloid leukemia (CBF AML) cell line treated with patient plasma.

CONTACTS AND LOCATIONS:
Overall Officials: Melinda Pauly, MD, Principal Investigator — Emory University